CLINICAL TRIAL: NCT00134056
Title: Phase III Study of Docetaxel and Atrasentan Versus Docetaxel and Placebo for Patients With Advanced Hormone Refractory Prostate Cancer
Brief Title: S0421, Docetaxel and Prednisone With or Without Atrasentan in Treating Patients With Stage IV Prostate Cancer and Bone Metastases That Did Not Respond to Previous Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000439434; S0421 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Atrasentan; Docetaxel; Prednisone; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: placebo (Active Comparator): Patients receive docetaxel and prednisone as in arm I. Patients also receive oral placebo once daily on days 1-21. Treatment repeat every 21 days for up to 12 courses. Patients with stable or responding disease after course 12 may register for continued oral placebo treatment for up to 52 weeks.
  Interventions: Drug: docetaxel; Drug: prednisone; Other: placebo
- Arm II: atrasentan hydrochloride (Experimental): Patients receive docetaxel IV over 1 hour on day 1. Patients also receive oral atrasentan and oral prednisone once daily on days 1-21. Treatment repeats every 21 days for up to 12 courses. Patients with stable or responding disease after course 12 may register for continued oral atrasentan treatment for up to 52 weeks.
  Interventions: Drug: atrasentan hydrochloride; Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: atrasentan hydrochloride — Given orally
  Other Names: atrasentan
  Arms: Arm II: atrasentan hydrochloride
Drug: docetaxel — Docetaxel given IV and prednisone given orally
  Other Names: taxotere
Drug: prednisone — Docetaxel given IV and prednisone given orally
  Other Names: steroid
Other: placebo — Given orally
  Arms: Arm I: placebo

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, prednisone, and atrasentan work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether docetaxel, prednisone, and atrasentan are more effective than docetaxel and prednisone in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying docetaxel, prednisone, and atrasentan to see how well they work compared to docetaxel and prednisone in treating patients with stage IV prostate cancer and bone metastases that did not respond to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival and progression-free survival of patients with hormone-refractory stage IV prostate cancer and bone metastases treated with docetaxel and prednisone combined with either atrasentan vs placebo.

Secondary

* Compare pain progression of patients treated with these regimens.
* Compare the qualitative and quantitative toxicity of these regimens in these patients.
* Compare the quality of life, in terms of palliation of metastatic bone pain and improvement in functional status, of patients treated with these regimens.
* Compare prostate-specific antigen (PSA) response rates in patients treated with these regimens.
* Compare objective response in patients with measurable disease treated with these regimens.
* Determine whether a 30% reduction in PSA and the slope of PSA from baseline to 3 months is a surrogate marker for survival in patients treated with these regimens.
* Correlate PSA progression with clinical progression and death in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease progression (measurable or non-measurable disease progression vs prostate-specific antigen progression only), use of bisphosphonates at study entry (yes vs no), worst pain, measured by the Brief Pain Inventory "pain" scale (< grade 4 vs ≥ grade 4), and extraskeletal metastases (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1. Patients also receive oral atrasentan and oral prednisone once daily on days 1-21. Treatment repeats every 21 days for up to 12 courses. Patients with stable or responding disease after course 12 may register for continued oral atrasentan treatment for up to 52 weeks in the absence of disease progression* or unacceptable toxicity.
* Arm II: Patients receive docetaxel and prednisone as in arm I. Patients also receive oral placebo once daily on days 1-21. Treatment repeat every 21 days for up to 12 courses. Patients with stable or responding disease after course 12 may register for continued oral placebo treatment for up to 52 weeks in the absence of disease progression* or unacceptable toxicity.

NOTE: *Patients with PSA progression alone will be allowed to continue treatment

Quality of life is assessed at baseline, before courses 4, 7, and 10, and then after completion of study treatment.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for up to 3 years from study entry.

PROJECTED ACCRUAL: A total of 930 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Stage IV disease (any T, any N, M1b)

    * Evidence of bone metastases by bone scan or MRI
* Measurable or nonmeasurable disease

  * Soft tissue disease that has been irradiated within the past 2 months is not assessable as measurable disease
* Hormone-refractory disease despite androgen deprivation and antiandrogen withdrawal, as defined by 1 of the following criteria:

  * Prostate-specific antigen (PSA) progression, defined as 3 consecutive rising PSA levels* taken ≥ 1 week apart

    * PSA ≥ 5 ng/mL NOTE: *If the third confirmatory PSA level is < the second level, the patient is considered eligible provided a fourth PSA level is > the second level
  * Progression of measurable disease
  * Progression of nonmeasurable disease by bone scan
* Must have undergone surgical or medical (e.g., luteinizing hormone-releasing hormone [LHRH] agonist [e.g., leuprolide or goserelin] or LHRH antagonist therapy) castration

  * Patients who have undergone medical castration must continue LHRH agonist or antagonist therapy during study treatment
* Must have completed 12 courses of blinding protocol treatment (atrasentan/placebo) AND stopped docetaxel for any reason (including completion of 12 courses) other than progressive disease
* No symptomatic pleural effusion
* No third space fluid accumulation (e.g., ascites)
* No prior or concurrent brain metastases

  * Patients with clinical evidence of brain metastases must have a negative brain CT scan or MRI within the past 8 weeks

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-3* NOTE: For a performance status of 3, the cause must be due to pain secondary to bone metastases

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Fertile patients must use effective contraception
* Able to take oral medication without crushing, dissolving, or chewing tablets
* No major infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II cancer in complete remission
* No symptomatic sensory neuropathy ≥ grade 2
* No history of hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No other significant, active medical illness that would preclude study treatment or survival

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 1 prior systemic vaccine or biologic therapy

  * At least 4 weeks since prior vaccine or biologic therapy and recovered
* No concurrent biological response modifiers
* No concurrent prophylactic colony-stimulating factors

Chemotherapy

* More than 2 years since prior adjuvant therapy with a single non-taxane-containing cytotoxic regimen
* No prior cytotoxic chemotherapy for metastatic prostate cancer
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 6 weeks since prior bicalutamide or nilutamide AND has subsequent disease progression
* At least 4 weeks since prior flutamide or ketoconazole AND has subsequent disease progression
* Prior or concurrent megestrol for treatment of hot flashes allowed
* No other concurrent corticosteroid or hormonal therapy unless continuing luteinizing hormone-releasing hormone treatment and/or bisphosphonate therapy

Radiotherapy

* See Disease Characteristics
* Prior samarium allowed
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to ≥ 30% of the bone marrow
* No prior strontium
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 3 weeks since prior surgery and recovered

Other

* More than 4 weeks since prior investigational drugs
* Concurrent bisphosphonates allowed provided therapy is started prior to study entry, dose is maintained during the first 12 weeks of study treatment, and patient meets criteria for disease progression

  * No initiation of bisphosphonates during the first 12 weeks of study treatment
* No concurrent herbal medications or food supplements (e.g., PC-SPES, saw palmetto, Hypericum perforatum [St. John's wort])

  * Concurrent daily vitamins and calcium supplements allowed
* At least 14 days since prior and no concurrent administration of any of the following:

  * Antibiotics (e.g., clarithromycin, erythromycin, troleandomycin, rifampin, rifabutin, and rifapentine)
  * Antifungals (e.g., itraconazole, ketoconazole, fluconazole [doses > 200 mg/day], and voriconazole)
  * Antidepressants (e.g., nefazodone and fluvoxamine)
  * Calcium channel blockers (e.g., verapamil, diltiazem)
  * Miscellaneous (e.g., amiodarone [no use within 6 months prior to study entry], grapefruit juice, bitter orange, or modafinil)
  * Anticonvulsants (e.g., phenytoin, carbamazepine, phenobarbital, and oxcarbazepine)
  * Antibiotics (e.g., rifampin, rifabutin, and rifapentine)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1038 (Actual)
Dates: Start 2006-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David I. Quinn, MD, Study Chair — University of Southern California; Maha Hadi A. Hussain, MD, Study Chair — University of Michigan Rogel Cancer Center; Primo N. Lara, MD, Study Chair — University of California, Davis; Mark Garzotto, MD, Study Chair — Portland VA Medical Center
Locations (554):
- United States (554):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Valley Medical Oncology, Fremont, California
  - Cancer Care Associates, Fresno, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Community Hospital of the Monterey Peninsula Comprehensive Cancer Center, Monterey, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - PCR Oncology, Pismo Beach, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Lucy Curci Cancer Center at Eisenhower Memorial Hospital and Medical Center, Rancho Mirage, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Connecticut Oncology & Hematology - Torrington, Torrington, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Cancer Centers of Central Florida, PA, Leesburg, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Space Coast Medical Associates, Titusville, Florida
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Leonard C. Ferguson Cancer Center, Freeport, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Central Dupage Cancer Center, Winfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Bloomington Hospital Regional Cancer Institute, Bloomington, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Medical Consultants, PC at Ball Memorial Cancer Center, Muncie, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - MetroWest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Frontier Cancer Center, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Riverside Middle Peninsula Cancer Center, Gloucester, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Peninsula Cancer Institute - Newport News Office, Newport News, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Peninsula Cancer Institute - Williamsburg Office, Williamsburg, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Oncology Alliance - Franklin, Franklin, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Oncology Alliance - Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Oncology Alliance, SC - Milwaukee - South, Milwaukee, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
http://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Result] Goldkorn A, Ely B, Quinn DI, et al.: Results of telomerase activity measurements from live circulating tumor cells captured on a slot microfilter in a phase III SWOG-coordinated prostate cancer trial (S0421). [Abstract] J Clin Oncol 30 (Suppl 15): A-4663, 2012.
- [Result] Lara P, Ely B, Quinn DI, et al.: SWOG 0421: prognostic and predictive value of bone metabolism biomarkers (BMB) in castration resistant prostate cancer (CRPC) patients (pts) with skeletal metastases treated with docetaxel (DOC) with or without atrasentan (ATR). [Abstract] J Clin Oncol 30 (Suppl 15): A-4547, 2012.
- [Result] Quinn DI, Tangen CM, Hussain M, et al.: SWOG S0421: phase III study of docetaxel (D) and atrasentan (A) versus docetaxel and placebo (P) for men with advanced castrate resistant prostate cancer (CRPC). [Abstract] J Clin Oncol 30 (Suppl 15): A-4511, 2012.
- [Result] Goldkorn A, Ely B, Quinn DI, Tangen CM, Fink LM, Xu T, Twardowski P, Van Veldhuizen PJ, Agarwal N, Carducci MA, Monk JP 3rd, Datar RH, Garzotto M, Mack PC, Lara P Jr, Higano CS, Hussain M, Thompson IM Jr, Cote RJ, Vogelzang NJ. Circulating tumor cell counts are prognostic of overall survival in SWOG S0421: a phase III trial of docetaxel with or without atrasentan for metastatic castration-resistant prostate cancer. J Clin Oncol. 2014 Apr 10;32(11):1136-42. doi: 10.1200/JCO.2013.51.7417. Epub 2014 Mar 10. PMID 24616308
- [Result] Goldkorn A, Xu T, Lu B, et al.: Circulating tumor cell capture and analysis in a multicenter SWOG-coordinated prostate cancer trial. [Abstract] J Clin Oncol 28 (Suppl 15): A-TPS342, 2010.
- [Derived] Lara PN Jr, Ely B, Quinn DI, Mack PC, Tangen C, Gertz E, Twardowski PW, Goldkorn A, Hussain M, Vogelzang NJ, Thompson IM, Van Loan MD. Serum biomarkers of bone metabolism in castration-resistant prostate cancer patients with skeletal metastases: results from SWOG 0421. J Natl Cancer Inst. 2014 Apr;106(4):dju013. doi: 10.1093/jnci/dju013. Epub 2014 Feb 24. PMID 24565955
- [Derived] Quinn DI, Tangen CM, Hussain M, Lara PN Jr, Goldkorn A, Moinpour CM, Garzotto MG, Mack PC, Carducci MA, Monk JP, Twardowski PW, Van Veldhuizen PJ, Agarwal N, Higano CS, Vogelzang NJ, Thompson IM Jr. Docetaxel and atrasentan versus docetaxel and placebo for men with advanced castration-resistant prostate cancer (SWOG S0421): a randomised phase 3 trial. Lancet Oncol. 2013 Aug;14(9):893-900. doi: 10.1016/S1470-2045(13)70294-8. Epub 2013 Jul 17. PMID 23871417
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II: Atrasentan: Patients receive docetaxel IV over 1 hour on day 1. Patients also receive oral atrasentan and oral prednisone once daily on days 1-21. Treatment repeats every 21 days for up to 12 courses. Patients with stable or responding disease after course 12 may register for continued oral atrasentan treatment for up to 52 weeks.
  atrasentan hydrochloride: Given orally
  docetaxel: Docetaxel given IV and prednisone given orally
  prednisone: Docetaxel given IV and prednisone given orally
Period: Randomization
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Started | 518 | 520
Completed | 496 | 500
Not Completed | 22 | 20
Not completed — Not eligible for assigned treatment | 22 | 20
Period: Eligible for Protocol Assigned Treatment
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Started | 496 | 500
Completed | 169 | 185
Not Completed | 327 | 315
Not completed — Lack of Efficacy | 171 | 171
Not completed — Adverse Event | 81 | 67
Not completed — Withdrawal by Subject | 20 | 21
Not completed — Other | 55 | 56

BASELINE CHARACTERISTICS:
Population: A total of 1038 patients were randomized to this study, 42 of which were ineligible. Baseline analysis population includes 994 patients (excluding the 42 ineligible patients and 2 additional patients who withdrew all consent prior to receiving protocol treatment).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Placebo | Arm II: Atrasentan | Total
Number analyzed (Participants) | 496 | 498 | 994
Age, Continuous [Median (Full Range); unit: years] | 69 [43 to 89] | 69 [40 to 92] | 69 [40 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 496 | 498 | 994
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 21 | 41
  Not Hispanic or Latino | 476 | 477 | 953
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 403 | 403 | 806
  Black | 64 | 73 | 137
  Asian | 12 | 8 | 20
  Unknown | 14 | 10 | 24
Serum PSA [Median (Inter-Quartile Range); unit: ug/L] | 67.7 [24.6 to 202.4] | 79.0 [23.5 to 228.3] | 72.7 [24.4 to 213.8]
Type of Progression at study entry [Count of Participants; unit: Participants]
  Measurable or evaluable | 394 | 407 | 801
  PSA increase only | 102 | 91 | 193
Bisphosphonate use at study entry [Count of Participants; unit: Participants] | 305 | 304 | 609
Brief Pain Inventory, worst pain [Count of Participants; unit: Participants] — score >=4 vs <4 in the Brief Pain Inventory scale for worst pain
  Participants
    >= 4 | 213 | 210 | 423
    <4 | 283 | 288 | 571
Metastases [Count of Participants; unit: Participants]
  Skeletal only | 206 | 203 | 409
  Lymph nodes | 148 | 149 | 297
  Lung, liver or brain | 94 | 101 | 195
  Extraskeletal | 48 | 45 | 93
Previous prostatectomy [Count of Participants; unit: Participants] | 145 | 168 | 313
Performance status [Count of Participants; unit: Participants] — SWOG Performance status:
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. = Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. = Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  Participants
    2-3 | 39 | 36 | 75
    0-1 | 457 | 462 | 919
Gleason score [Count of Participants; unit: Participants] — Pathologists grade prostate cancers using numbers from 1 to 5 based on how much the cells in the cancerous tissue look like normal tissue. This is called the Gleason system.
  If the cancerous tissue looks like normal tissue, a grade of 1 is assigned. If the cancer cells look very abnormal, a grade of 5 is assigned. Grades 2-4 have features in between these extremes.
  Since prostate cancers often have areas with different grades, a grade is assigned to the 2 areas that make up most of the cancer. These 2 grades are added to yield the Gleason score. The highest a Gleason score can be is 10.
  Participants
    5-6 | 49 | 52 | 101
    7 | 137 | 141 | 278
    8-10 | 272 | 275 | 547
    Missing | 38 | 30 | 68

OUTCOME MEASURES:

1. Primary Outcome: Compare Survival Between a Control or Standard Therapy Arm of Docetaxel + Placebo + Prednisone With Docetaxel + Atrasentan + Prednisone in Patients With Hormone Refractory Prostate Cancer.
Description: Measured from date of registration to date of death due to any cause. Patient last known to be alive are censored at date of last contact.
Time Frame: Up to 7 years after study opens
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Number analyzed (Participants) | 496 | 498
months | 17.6 [16.4 to 20.1] | 17.8 [16.4 to 19.8]
Statistical Analysis 1: Comparison: Arm I: Placebo vs Arm II: Atrasentan; The primary analysis was by intention to treat and the Hochberg procedure was used for multiple testing of co-primary endpoints. Assuming a 4 year accrual, 2.5 years of follow-up, and 930 eligible patients, the study was designed to have 87% power to detect a 25% increase from 18.0 months to 22.5 months in median overall survival with a one-sided log rank with alpha of 0.0125; Test type: Superiority or Other; p = 0.64, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.90 to 1.19]

2. Primary Outcome: Compare Progression-free Survival Between a Control or Standard Therapy Arm of Docetaxel + Placebo + Prednisone With Docetaxel + Atrasentan + Prednisone in Patients With Hormone Refractory Prostate Cancer.
Description: Measured from date of registration to date of first observation of progressive disease, or death due to any cause. Patients without progression are censored at date of last contact. Disease progression is defined by confirmed bone disease progression, soft tissue or pain progression.
Time Frame: Up to 7 years after study opens
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Number analyzed (Participants) | 496 | 498
months | 9.1 [8.4 to 10.2] | 9.2 [8.5 to 9.9]
Statistical Analysis 1: Comparison: Arm I: Placebo vs Arm II: Atrasentan; The primary analysis was by intention to treat and the Hochberg procedure was used for multiple testing of co-primary endpoints. Assuming a 4 year accrual, 2.5 years of follow-up, and 930 eligible patients, the study was designed to have 87% power to detect a 25% increase from 6.0 months to 7.5 months in median overall survival with a one-sided log rank with alpha of 0.0125; Test type: Superiority or Other; p = 0.81, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.89 to 1.16]

3. Secondary Outcome: Compare Pain Progression Between the Two Study Arms.
Description: Pain progression is defined as patients reporting an increase of at least two Worst Pain points, maintained for at least two consecutive assessments, increase to Level 3 (strong opioid) on the Pain Medication Log Analgesic Code for patients receiving Level 2 (weak opioid) analgesics at randomization, or an increase to Level 2 or 3 analgesics for patients receiving Level 0 or 1 analgesics at randomization.
Time Frame: Up to 52 weeks
Population: Only those patients who progressed on study were included in this analysis. The proportion of patients with pain progression is calculated using number of patients with pain progression as the numerator and the total number of patients who progressed on study as the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Number analyzed (Participants) | 416 | 408
Participants | 59 | 41

4. Secondary Outcome: Compare Qualitative and Quantitative Toxicity Between the Two Study Arms
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Assessed every 3 weeks up to 52 weeks
Population: patients with hormone-refractory stage IV prostate cancer and bone metastases treated with docetaxel and prednisone combined with either atrasentan vs placebo
Measure: Number; unit: Participants
Groups:
- Arm II: Atrasentan: Patients receive docetaxel IV over 1 hour on day 1. Patients also receive oral atrasentan and oral prednisone once daily on days 1-21. Treatment repeats every 21 days for up to 12 courses. Patients with stable or responding disease after course 12 may register for continued oral atrasentan treatment for up to 52 weeks.
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Number analyzed (Participants) | 486 | 492
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 2 | 2
  AST, SGOT | 2 | 4
  Adult respiratory distress syndrome (ARDS) | 3 | 0
  Albumin, serum-low (hypoalbuminemia) | 3 | 0
  Alkaline phosphatase | 4 | 6
  Allergic reaction/hypersensitivity | 5 | 6
  Allergy/Immunology-Other (Specify) | 0 | 1
  Amylase | 0 | 1
  Anorexia | 5 | 5
  Arthritis (non-septic) | 1 | 0
  Aspiration | 0 | 1
  Auditory/Ear-Other (Specify) | 1 | 0
  Bilirubin (hyperbilirubinemia) | 0 | 1
  Blood/Bone Marrow-Other (Specify) | 2 | 2
  CNS cerebrovascular ischemia | 0 | 1
  CPK (creatine phosphokinase) | 2 | 0
  Calcium, serum-low (hypocalcemia) | 7 | 1
  Cardiac Arrhythmia-Other (Specify) | 2 | 0
  Cardiac General-Other (Specify) | 1 | 1
  Cardiac troponin I (cTnI) | 2 | 1
  Cardiac troponin T (cTnT) | 1 | 0
  Cardiac-ischemia/infarction | 2 | 1
  Conduction abnormality NOS | 1 | 0
  Confusion | 1 | 0
  Constipation | 3 | 4
  Cough | 1 | 2
  Creatinine | 4 | 1
  Dehydration | 9 | 8
  Diarrhea | 10 | 7
  Dizziness | 3 | 1
  Dry mouth/salivary gland (xerostomia) | 1 | 0
  Dysphagia (difficulty swallowing) | 1 | 1
  Dyspnea (shortness of breath) | 38 | 17
  Edema: head and neck | 0 | 1
  Edema: limb | 16 | 2
  Edema: trunk/genital | 1 | 0
  Erectile dysfunction | 2 | 0
  Esophagitis | 0 | 1
  Fatigue (asthenia, lethargy, malaise) | 60 | 40
  Febrile neutropenia | 8 | 20
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 1 | 2
  Fracture | 1 | 0
  Glucose, serum-high (hyperglycemia) | 20 | 24
  Glucose, serum-low (hypoglycemia) | 1 | 0
  Heartburn/dyspepsia | 1 | 1
  Hemoglobin | 47 | 22
  Hemolysis | 1 | 0
  Hemorrhage, Respiratory tract NOS | 0 | 1
  Hemorrhage, GI - Rectum | 1 | 0
  Hemorrhage, GI - Stomach | 1 | 0
  Hemorrhage, GI - Upper GI NOS | 0 | 1
  Hemorrhage, GU - Bladder | 0 | 1
  Hemorrhage/Bleeding-Other (Specify) | 2 | 1
  Hemorrhoids | 0 | 2
  Hot flashes/flushes | 2 | 1
  Hypertension | 2 | 2
  Hypotension | 9 | 3
  Hypoxia | 10 | 3
  INR (of prothrombin time) | 3 | 1
  Induration/fibrosis (skin and subcutaneous tissue) | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Bladder | 1 | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 2 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Bronchus | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Esophagus | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 11 | 6
  Inf (clin/microbio) w/Gr 3-4 neuts - Nerve-periph | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1 | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Soft tissue | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 4 | 3
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 0 | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus | 1 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Colon | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1 | 5
  Inf w/normal ANC or Gr 1-2 neutrophils - Muscle | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Scrotum | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Sinus | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 1 | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Stomach | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Trachea | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Ungual | 0 | 1
  Inf w/unknown ANC - Middle ear (otitis media) | 0 | 1
  Inf w/unknown ANC - Upper aerodigestive NOS | 0 | 1
  Infection with unknown ANC - Blood | 0 | 1
  Infection with unknown ANC - Lung (pneumonia) | 3 | 0
  Infection with unknown ANC - Upper airway NOS | 0 | 1
  Infection with unknown ANC - Urinary tract NOS | 1 | 1
  Infection-Other (Specify) | 4 | 3
  Insomnia | 1 | 1
  Left ventricular diastolic dysfunction | 1 | 0
  Left ventricular systolic dysfunction | 3 | 2
  Leukocytes (total WBC) | 101 | 98
  Lipase | 0 | 1
  Lymphopenia | 30 | 32
  Magnesium, serum-high (hypermagnesemia) | 1 | 0
  Metabolic/Laboratory-Other (Specify) | 0 | 2
  Mood alteration - agitation | 1 | 0
  Mood alteration - depression | 1 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 2 | 2
  Mucositis/stomatitis (clinical exam) - Pharynx | 1 | 0
  Mucositis/stomatitis (clinical exam) - Stomach | 1 | 0
  Mucositis/stomatitis (functional/symp) - Esophagus | 0 | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 3 | 3
  Mucositis/stomatitis (functional/symp) - Pharynx | 0 | 1
  Mucositis/stomatitis (functional/symp) - Rectum | 0 | 1
  Muscle weakness, not d/t neuropathy - Extrem-lower | 2 | 1
  Muscle weakness, not d/t neuropathy - body/general | 11 | 8
  Myocarditis | 1 | 0
  Nail changes | 0 | 1
  Nasal cavity/paranasal sinus reactions | 2 | 0
  Nausea | 11 | 5
  Neuropathy: motor | 7 | 6
  Neuropathy: sensory | 10 | 11
  Neutrophils/granulocytes (ANC/AGC) | 140 | 154
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 1 | 1
  PTT (Partial thromboplastin time) | 1 | 0
  Pain - Abdomen NOS | 4 | 0
  Pain - Back | 1 | 2
  Pain - Bone | 5 | 8
  Pain - Chest wall | 0 | 1
  Pain - Chest/thorax NOS | 1 | 0
  Pain - Extremity-limb | 1 | 1
  Pain - Joint | 2 | 2
  Pain - Muscle | 8 | 3
  Pain - Neuralgia/peripheral nerve | 1 | 1
  Pain - Pelvis | 0 | 1
  Pain-Other (Specify) | 0 | 1
  Phosphate, serum-low (hypophosphatemia) | 3 | 0
  Platelets | 7 | 4
  Pneumonitis/pulmonary infiltrates | 7 | 0
  Pneumothorax | 1 | 0
  Potassium, serum-high (hyperkalemia) | 2 | 1
  Potassium, serum-low (hypokalemia) | 11 | 2
  Pulmonary/Upper Respiratory-Other (Specify) | 0 | 1
  Rash: hand-foot skin reaction | 1 | 0
  Renal failure | 4 | 2
  Renal/Genitourinary-Other (Specify) | 1 | 0
  Right ventricular dysfunction (cor pulmonale) | 0 | 1
  SVT and nodal arrhythmia - Atrial fibrillation | 3 | 2
  SVT and nodal arrhythmia - Atrial flutter | 1 | 1
  SVT and nodal arrhythmia - Sinus tachycardia | 0 | 1
  Sodium, serum-low (hyponatremia) | 8 | 3
  Somnolence/depressed level of consciousness | 1 | 0
  Speech impairment (e.g., dysphasia or aphasia) | 0 | 1
  Sudden death | 2 | 0
  Syncope (fainting) | 3 | 1
  Thrombosis/embolism (vascular access-related) | 0 | 1
  Thrombosis/thrombus/embolism | 9 | 11
  Vasovagal episode | 0 | 2
  Vomiting | 8 | 7
  Watery eye (epiphora, tearing) | 0 | 1
  Weight gain | 0 | 1

5. Secondary Outcome: Compare Prostate Specific Antigen (PSA) Response Rates Between the Experimental Arm and the Standard Arm.
Description: PSA Partial Response: Greater than or equal to 50% reduction in baseline PSA. There must be no evidence of soft tissue progression, or confirmed none disease progression, or pain progression.
Time Frame: Up to 7 years after study opens
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Number analyzed (Participants) | 496 | 498
Participants | 243 | 249

6. Secondary Outcome: Compare Objective Responses Between the Two Treatment Groups in Patients With Measurable Disease as Defined by RECIST Criteria.
Description: Complete Response (CR): Complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. Normalization of markers and other abnormal lab values. PSA ≤ .2 ng/ml. Partial Response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions.
Time Frame: Up to 52 weeks
Population: 450 (225 in each arm) of 461 patients with measurable disease at trial enrollment were assessable for response by RECIST.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Number analyzed (Participants) | 225 | 225
Participants
  Partial response (confirmed) | 31 | 32
  Complete response | 0 | 0
  No response | 194 | 193

7. Other Pre Specified Outcome: Compare Elements of Quality of Life Between Treatment Arms: Pain Palliation Response, as Measured by the Brief Pain Inventory (BPI)
Description: Pain palliation is the proportion of patients showing a two-point reduction in the Worst Pain score (WPS) maintained for two consecutive assessments with no increase in analgesic use. Increase in analgesic use is defined as an increase in Analgesic code Level to 2 (weak opioid) or 3 (strong opioid). Patients will be classified as pain palliated or not palliated. Patients with a WPS of "0" will be defined as "stable" if their WPS remains "0" for Weeks 7 and 10 with no increase in analgesic use, but they will not be categorized as responders. Pain palliation response is measured by BPI short form that has the following: yes/no question about pain today; 4 pain rating questions (worst pain, least pain, average pain, and current pain); pain medications and pain relief; 7 items addressing effect of pain on functioning. For patients who continue to receive treatment beyond 12 treatment cycles, the Worst Pain item is measured by Pain Medication Log and Pain Assessment
Time Frame: up to 18 months study period
Population: There was a large amount of missing data points due to the difficulty of data collection of pain medication logs in addition to a questionnaire.The study team and site staff were only able to obtain complete data for the patients included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Number analyzed (Participants) | 274 | 260
Participants | 75 | 83

8. Other Pre Specified Outcome: Number of Patients With a Change in Functional Status
Description: Functional status will be measured with the Functional Assessment of Cancer Therapy-Prostate (FACT-P) Trial Outcome Index. The FACT-P also addresses four general domains of QOL (physical, functional, emotional, and social well-being subscales) as well as symptom concerns associated with prostate cancer and its treatment.
Time Frame: up to 18 months study period
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Placebo | Arm II: Atrasentan Hydrochloride
Number analyzed (Participants) | 487 | 484
Participants | 118 | 139

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks up to 52 weeks
Description: Participants were monitored for toxicity every 3 weeks while on protocol therapy or at more frequent intervals appropriate for that participant, as judged by the treating physician.
Arm/Group | Arm I: Placebo | Arm II: Atrasentan
Serious Adverse Events (participants affected / at risk) | 172/486 | 153/492
Other Adverse Events (participants affected / at risk) | 476/486 | 475/492
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Placebo (N=486) | Arm II: Atrasentan (N=492)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 9
Hemoglobin (Blood and lymphatic system disorders) | 10 | 5
Cardiac General-Other (Cardiac disorders) | 3 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 7 | 2
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 0 | 2
Left ventricular diastolic dysfunction (Cardiac disorders) | 2 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 2
Myocarditis (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (cor pulmonale) (Cardiac disorders) | 0 | 1
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 8 | 3
SVT and nodal arrhythmia - Atrial flutter (Cardiac disorders) | 3 | 2
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia - PVCs (Cardiac disorders) | 1 | 0
Ventricular arrhythmia - Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 1 | 0
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1 | 0
Vision-blurred vision (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 4
Distention/bloating, abdominal (Gastrointestinal disorders) | 1 | 0
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal-Other (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Abdomen NOS (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 1 | 1
Hemorrhage, GI - Duodenum (Gastrointestinal disorders) | 2 | 2
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 0 | 1
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 3 | 2
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1 | 3
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 1 | 0
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 0 | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 5 | 6
Obstruction, GI - Colon (Gastrointestinal disorders) | 0 | 1
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 3
Pain - Abdomen NOS (Gastrointestinal disorders) | 7 | 5
Perforation, GI - Colon (Gastrointestinal disorders) | 1 | 0
Perforation, GI - Duodenum (Gastrointestinal disorders) | 0 | 1
Perforation, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Stricture/stenosis (including anastomotic), GI - A (Gastrointestinal disorders) | 1 | 0
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 2 | 2
Ulcer, GI - Rectum (Gastrointestinal disorders) | 1 | 0
Ulcer, GI - Stomach (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 9
Death - Multi-organ failure (General disorders) | 3 | 0
Death not associated with CTCAE term - Death NOS (General disorders) | 4 | 5
Edema: head and neck (General disorders) | 0 | 1
Edema: limb (General disorders) | 4 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14 | 6
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 0 | 1
Pain - Chest/thorax NOS (General disorders) | 2 | 2
Pain - Pain NOS (General disorders) | 0 | 1
Pain-Other (General disorders) | 3 | 1
Sudden death (General disorders) | 3 | 2
Inf (clin/microbio) w/Gr 3-4 neuts - Appendix (Infections and infestations) | 0 | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Bladder (Infections and infestations) | 1 | 2
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 4 | 3
Inf (clin/microbio) w/Gr 3-4 neuts - Colon (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Eye NOS (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 14 | 8
Inf (clin/microbio) w/Gr 3-4 neuts - Nerve-periph (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Nose (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Pharynx (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - UTI (Infections and infestations) | 7 | 6
Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Ab NOS (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bladder (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 5 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Catheter (Infections and infestations) | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Colon (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Liver (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 12 | 9
Inf w/normal ANC or Gr 1-2 neutrophils - Mid ear (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Muscle (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Scrotum (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 3 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Trachea (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 3 | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Wound (Infections and infestations) | 0 | 2
Inf w/normal ANC or Gr 1-2 neutrophils -Nerve-peri (Infections and infestations) | 0 | 1
Inf w/unknown ANC - Middle ear (otitis media) (Infections and infestations) | 0 | 1
Inf w/unknown ANC - Upper aerodigestive NOS (Infections and infestations) | 0 | 1
Infection (documented clinically or microbiologica (Infections and infestations) | 2 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 0 | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 | 0
Infection with unknown ANC - Rectum (Infections and infestations) | 0 | 1
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 0 | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 | 1
Infection with unknown ANC - Wound (Infections and infestations) | 1 | 0
Infection-Other (Infections and infestations) | 1 | 1
Perforation, GI - Appendix (Infections and infestations) | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 5 | 3
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 1
AST, SGOT (Investigations) | 1 | 1
Alkaline phosphatase (Investigations) | 1 | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1 | 0
CPK (creatine phosphokinase) (Investigations) | 1 | 0
Cardiac troponin I (cTnI) (Investigations) | 5 | 1
Cardiac troponin T (cTnT) (Investigations) | 1 | 0
Creatinine (Investigations) | 6 | 4
Fibrinogen (Investigations) | 1 | 0
INR (of prothrombin time) (Investigations) | 1 | 1
Leukocytes (total WBC) (Investigations) | 8 | 8
Lymphopenia (Investigations) | 1 | 1
Metabolic/Laboratory-Other (Investigations) | 0 | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 15 | 11
Platelets (Investigations) | 1 | 0
Prolonged QTc interval (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 4
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 | 0
Dehydration (Metabolism and nutrition disorders) | 13 | 7
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 | 7
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 | 0
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 4
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain - Bone (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 11
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 1 | 3
Hemorrhage, CNS (Nervous system disorders) | 1 | 1
Mental status (Nervous system disorders) | 0 | 1
Neurology-Other (Nervous system disorders) | 0 | 1
Neuropathy: CN III Pupil, eyelid, xtra ocular mvmt (Nervous system disorders) | 0 | 1
Neuropathy: CN VII Motor-face; Sensory-taste (Nervous system disorders) | 0 | 1
Neuropathy: cranial - CN VI Lateral deviation of e (Nervous system disorders) | 0 | 1
Neuropathy: motor (Nervous system disorders) | 1 | 2
Pain - Head/headache (Nervous system disorders) | 0 | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 | 0
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 | 1
Syncope (fainting) (Nervous system disorders) | 4 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 1 | 0
Vasovagal episode (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 4 | 4
Mood alteration - depression (Psychiatric disorders) | 0 | 2
Personality/behavioral (Psychiatric disorders) | 0 | 1
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 | 1
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 0 | 2
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 | 1
Obstruction, GU - Ureter (Renal and urinary disorders) | 0 | 2
Obstruction, GU - Urethra (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 8 | 7
Renal/Genitourinary-Other (Renal and urinary disorders) | 1 | 0
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 3 | 3
Pain - Testicle (Reproductive system and breast disorders) | 0 | 1
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 25 | 9
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pulmonary fibrosis (radiographic changes) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 1 | 0
Pain - Scalp (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 13 | 7
Thrombosis/thrombus/embolism (Vascular disorders) | 12 | 17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Placebo (N=486) | Arm II: Atrasentan (N=492)
Hemoglobin (Blood and lymphatic system disorders) | 350 | 331
Vision-blurred vision (Eye disorders) | 26 | 14
Watery eye (epiphora, tearing) (Eye disorders) | 37 | 41
Constipation (Gastrointestinal disorders) | 185 | 176
Diarrhea (Gastrointestinal disorders) | 143 | 149
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 33 | 23
Heartburn/dyspepsia (Gastrointestinal disorders) | 36 | 43
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 39 | 27
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 30 | 46
Nausea (Gastrointestinal disorders) | 201 | 188
Pain - Abdomen NOS (Gastrointestinal disorders) | 29 | 46
Vomiting (Gastrointestinal disorders) | 78 | 62
Edema: limb (General disorders) | 284 | 178
Fatigue (asthenia, lethargy, malaise) (General disorders) | 357 | 346
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 43 | 30
Pain-Other (General disorders) | 32 | 34
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 27 | 21
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 33 | 36
AST, SGOT (Investigations) | 71 | 80
Alkaline phosphatase (Investigations) | 106 | 113
Creatinine (Investigations) | 79 | 71
Leukocytes (total WBC) (Investigations) | 165 | 165
Lymphopenia (Investigations) | 76 | 72
Metabolic/Laboratory-Other (Investigations) | 23 | 27
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 179 | 180
Platelets (Investigations) | 71 | 47
Weight gain (Investigations) | 49 | 36
Weight loss (Investigations) | 39 | 36
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 91 | 90
Anorexia (Metabolism and nutrition disorders) | 112 | 106
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 109 | 75
Dehydration (Metabolism and nutrition disorders) | 27 | 29
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 191 | 202
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 36 | 33
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 59 | 47
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 75 | 61
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 39 | 44
Pain - Back (Musculoskeletal and connective tissue disorders) | 85 | 86
Pain - Bone (Musculoskeletal and connective tissue disorders) | 138 | 156
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 41 | 45
Pain - Joint (Musculoskeletal and connective tissue disorders) | 112 | 119
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 119 | 104
Dizziness (Nervous system disorders) | 91 | 96
Neuropathy: motor (Nervous system disorders) | 25 | 43
Neuropathy: sensory (Nervous system disorders) | 202 | 223
Pain - Head/headache (Nervous system disorders) | 70 | 45
Taste alteration (dysgeusia) (Nervous system disorders) | 158 | 132
Insomnia (Psychiatric disorders) | 74 | 80
Mood alteration - anxiety (Psychiatric disorders) | 20 | 27
Mood alteration - depression (Psychiatric disorders) | 37 | 28
Urinary frequency/urgency (Renal and urinary disorders) | 48 | 58
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 78 | 50
Cough (Respiratory, thoracic and mediastinal disorders) | 92 | 80
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 197 | 156
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 17 | 29
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 40 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 28 | 33
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 201 | 192
Nail changes (Skin and subcutaneous tissue disorders) | 97 | 149
Rash/desquamation (Skin and subcutaneous tissue disorders) | 45 | 70
Hot flashes/flushes (Vascular disorders) | 65 | 71
Hypertension (Vascular disorders) | 14 | 35
Hypotension (Vascular disorders) | 69 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No